CLINICAL TRIAL: NCT03676933
Title: A Prospective, Randomised, Vehicle-Controlled, Double-Blind, Exploratory Clinical Trial To Assess The Efficacy And Steroid Sparing Potential Of DGLA Cream Topically Applied To Early Childhood Patients With Moderate To Severe Atopic Dermatitis
Brief Title: Efficacy and Steroid Sparing Potential Study of DGLA Cream in Early Childhood Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DS Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS107E-05
Record Dates: First submitted 2018-01-30; First posted 2018-09-19 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — hydrocortisone-17-butyrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS107E and Steroid (Experimental): First 7 days: Steroid taken topically once a day and DS107E taken once a day Next 56 days: DS107E taken topically twice a day
  Interventions: Drug: DS107E; Drug: Hydrocortisone Butyrate 0.1% Cream
- Vehicle and Steroid (Placebo Comparator): First 7 days: Steroid taken topically once a day and DS107E taken once a day Next 56 days: DS107E taken topically twice a day
  Interventions: Drug: Vehicle; Drug: Hydrocortisone Butyrate 0.1% Cream

INTERVENTIONS:
Drug: DS107E
  Arms: DS107E and Steroid
Drug: Vehicle
  Arms: Vehicle and Steroid
Drug: Hydrocortisone Butyrate 0.1% Cream — Steroid taken topically once a day

SUMMARY:
This study will investigate the steroid sparing potential of DS107E to vehicle in patients with moderate to severe atopic dermatitis.

DS107E or vehicle will be topically administered with a steroid twice a day for the first 7 days. For the following 56 days DS107E or vehicle will be topically administered twice a day.

This study will enrol approximately 40 paediatric patients.

DETAILED DESCRIPTION:
Patients will come to the clinic on 8 occasions: Screening, Baseline, Day 7, Day 21, Day 35, Day 49, Day 63 (End of Treatment) and Day 91 (Follow-up). The primary efficacy variables will be IGA (Investigator Global Assessment) and SCORAD (SCORing Atopic Dermatitis) .

The secondary efficacy variables will be IGA, SCORAD, EASI (Eczema Area and Severity Index), IDQOL (Infant Dermatology Quality of Life), DFI (Dermatitis Family Impact), BSA, TEWL (Transepidermal Water Loss) and Time to Rescue Medication.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male infants aged 3-12 months.
2. Diagnosis of atopic dermatitis according to the Hanifin and Rajka Criteria.
3. Patients with moderate to severe atopic dermatitis (IGA ≥3)
4. Patients with atopic dermatitis covering a minimum of 10% of the body surface area at baseline.
5. Atopic Dermatitis is stable for the past 7 days, in the opinion of the investigator.
6. The patient's parents are able to apply the study product twice a day (each morning and evening) for a consecutive period of 63 days.
7. Patients who have completed the tolerability patch test without any adverse effects after 72 hours.

Exclusion Criteria:

1. Any clinically significant controlled or uncontrolled medical condition that would, in the opinion of the investigator, put the patient at undue risk or interfere with interpretation of study results.
2. Clinically significant impairment of renal or hepatic function.
3. Clinically significant immunodeficiency.
4. Use of systemic antibiotics less than 2 weeks prior to Baseline Visit (Day 0).
5. Other skin conditions that might interfere with atopic dermatitis diagnosis and/or evaluation (such as psoriasis or current viral, bacterial and fungal skin infections).
6. History of intolerance to any ingredient in DS107E DGLA cream or Vehicle cream (including the tolerability patch test performed at the Screening Visit) or intolerance to any ingredient in Locoid® Ointment (hydrocortisone butyrate 0.1%).
7. Use of systemic treatments that could affect atopic dermatitis less than 4 weeks prior to Baseline Visit (Day 0), e.g. oral corticosteroids; Intranasal corticosteroids and inhaled corticosteroids for stable medical conditions are allowed.
8. Treatment with any experimental drug within 30 days prior to Day 0 Visit (Baseline), or 5 half-lives (whichever is longer).
9. Excessive sun exposure or other ultraviolet (UV) light sources 4 weeks prior to Day 0 Visit (Baseline) and/or is planning a trip to sunny climate or other UV sources between screening and follow-up visits.
10. Use of any topical medicated treatment for atopic dermatitis 2 weeks prior to start of treatment/Day 0 Visit (Baseline), including but not limited to topical corticosteroids, calcineurin inhibitors, tars, bleach, antimicrobials and bleach baths.
11. Use of topical products containing ceramides 2 weeks prior to Day 0.
12. Medical history of chronic infectious disease (e.g., hepatitis B, hepatitis C or infection with human immunodeficiency virus).

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04-25 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | 9 weeks
SCORing Atopic Dermatitis | 9 weeks
  Erythema, population, oozing, excoriation, lichenification, dryness, body surface area, sleep loss and pruritus is all graded. The sum of the above measures represent the SCORAD which can vary from 0 to 103.

SECONDARY OUTCOMES:
Investigator Global Assessment | Days 7, 21. 35. 49, 63
Eczema Area and Severity Index | Days 7, 21. 35. 49, 63
  Proportion of patients achieving a reduction in EASI score
Body Surface Area | Days 7, 21. 35. 49, 63
Trans-Epidermal Water Loss | Days 63
Time to Rescue Medication | 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- DS Biopharma Investigational Site, Dublin, Ireland